CLINICAL TRIAL: NCT05768230
Title: Using Transesophageal Echocardiography to Evaluate the Effect of Levosimendan on Patients With Acute Respiratory Distress Syndrome Associated With Right Ventricular Dysfunction During Mechanical Ventilation
Brief Title: Using TEE to Evaluate the Effect of Levosimendan on Patients With ARDS Associated With RVD During MV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARVD20220810
Record Dates: First submitted 2023-02-18; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-12

CONDITIONS: Transesophageal Echocardiography; Acute Respiratory Distress Syndrome; Right Ventricular Dysfunction
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventricular Dysfunction, Right | interventions — Simendan; Glucose

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to treatment group A: intravenously injected levosimendan 12.5mg with 5% glucose injection 50ml configuration at 2ml/h for 24h, or treatment group B: control group with 5% glucose injection 2ml/h for 24h.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group A (Experimental): intravenously injected levosimendan 12.5mg with 5% glucose injection 50ml configuration at 2ml/h for 24h
  Interventions: Drug: levosimendan
- treatment group B (Placebo Comparator): treatment group B: control group with 5% glucose injection 2ml/h for 24h
  Interventions: Drug: 5% glucose injection

INTERVENTIONS:
Drug: levosimendan — Levosimendan 12.5mg was injected intravenously in a 5% glucose injection 50ml configuration at a rate of 2ml/h for 24 hours.The injection was performed at a constant rate of 2ml/h. If there was no significant hypotension or tachycardia, the injection was completed within 24h
  Arms: treatment group A
Drug: 5% glucose injection — 5% glucose injection 50ml configuration at a rate of 2ml/h for 24 hours.The injection was performed at a constant rate of 2ml/h. If there was no significant hypotension or tachycardia, the injection was completed within 24h
  Arms: treatment group B

SUMMARY:
Acute respiratory distress syndrome (ARDS) is often complicated by right ventricular dysfunction (RVD), Acute cor pulmonale is the most serious form of ARDS complicated with RVD.Levosimendan is indicated for short-term treatment of acute decompensated heart failure that is not responding well to conventional therapy and requires increased myocardial contractile force.In 2016, the European Society of Cardiology issued recommendations for the management of acute right heart failure, stating that levosimendan can improve right ventriculo-pulmonary artery coupling by both increasing right heart contractility and reducing pulmonary vascular resistance.However, the clinical application of levosimendan in the treatment of ARDS right heart dysfunction is insufficient.Therefore, this study intends to use transesophageal ultrasound to evaluate right ventricular function, reduce the limitation of poor right ventricular window in transthoracic echocardiography, and conduct a multi-center randomized controlled study to further explore the effects of levosimendan on right ventricular function in ARDS patients, such as tricuspid ring systolic displacement (TAPSE) and tricuspid ring systolic displacement velocity (S '). Effects of right ventricular area change fraction (RV FAC), right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA), pulmonary circulation resistance (PVR), hemodynamics and mortality.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is often complicated by right ventricular dysfunction (RVD),the incidence can be as high as 64%, Acute cor pulmonale is the most serious form of ARDS complicated with RVD. The prognosis of ARDS patients with RVD is worse and the risk of death would be significantly increased.Currently, there are very limited clinical drug treatment options for RVD.Levosimendan is indicated for short-term treatment of acute decompensated heart failure that is not responding well to conventional therapy and requires increased myocardial contractile force.In 2016, the European Society of Cardiology issued recommendations for the management of acute right heart failure, stating that levosimendan can improve right ventriculo-pulmonary artery coupling by both increasing right heart contractility and reducing pulmonary vascular resistance. Levosimendan is therefore recommended to be given priority over dobutamine in the treatment of acute right heart failure.At present, there are also relevant clinical studies reporting that levosimendan can be used in acute right heart failure caused by different causes, including a single center randomized controlled study reporting that levosimendan can do work in the right ventricle of patients with sepsis ARDS, and has beneficial hemodynamic effects.However, the clinical application of levosimendan in the treatment of ARDS right heart dysfunction is insufficient.Therefore, this study intends to use transesophageal ultrasound to evaluate right ventricular function, reduce the limitation of poor right ventricular window in transthoracic echocardiography, and conduct a multi-center randomized controlled study to further explore the effects of levosimendan on right ventricular function in ARDS patients, such as tricuspid ring systolic displacement (TAPSE) and tricuspid ring systolic displacement velocity (S '). Effects of right ventricular area change fraction (RV FAC), right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA), pulmonary circulation resistance (PVR), RV-PA coupling, hemodynamics and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in this clinical trial and sign informed consent
* Age 18-80 years old, gender unlimited
* Patients with ARDS(According to the diagnostic criteria of ARDS in Berlin 2012) requiring mechanical ventilation; Acute right ventricular dysfunction due to ARDS

Exclusion Criteria:

* Pregnant or lactating women;
* Chronic cardiac insufficiency, pulmonary hypertension and/or right ventricular enlargement caused by chronic cardiopulmonary disease, cardiogenic shock or after major cardiac surgery before ARDS;
* right ventricular myocardial infarction;
* Uncorrected hypotension, hypoxemia and hypercapnia, or acid-base balance disturbance
* Mechanical ventilation driving pressure >=18cmH2O before randomization
* Rapid arrhythmia;
* pericardial tamponade;
* Pulmonary embolism;
* severe renal insufficiency;
* severe liver insufficiency;
* Failure to sign informed consent;
* known allergy to the test drug and control drug;
* Patients who have participated in other clinical trials within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-22 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The rate of right ventricular dysfunction occurrence within 48 hours after randomization. | From the time point of enrollment to 48 hours after enrollment
  Right ventricular dysfunction(RVD) is diagnosed when the results of an echocardiogram show one of the following, including: tricuspid annular plane systolic excursion(TAPSE)<16 mm, right ventricular fractional area change(RV FAC)<35% or systolic velocity of the lateral tricuspid valve annulus( RV S')<10 cm/s.

SECONDARY OUTCOMES:
Right ventricular area fractional change (RV FAC) 48 hours after randomization | at the time of 48 hours after enrollment
  Right ventricular area fractional change (RV FAC)is a simple and repeatable ultrasound method for evaluating RV function. Methods: The RV end-diastolic area (RVEDA) and RV end-systolic area (RVESA) were measured on the apical four-chamber section by two-dimensional ultrasound. RV FAC=(RVEDA- RVESA)/RVEDA*100%.
tricuspid annular plane systolic excursion(TAPSE) 48 hours after randomization | at the time of 48 hours after enrollment
  TAPSE is one of the most effective ultrasound methods for evaluating right ventricular function.Measurement method: TAPSE was measured on the four-chamber section of the apex of the heart by M-mode ultrasound. the sampling line was placed at the side wall of the tricuspid valve ring, parallel to the free wall of the right ventricle as far as possible, and the displacement of the tricuspid valve ring was measured from the end of diastole to the end of systole.
Tricuspid annular systolic S' velocity (TS') | at the time of 48 hours after enrollment
  TS' is an objective and accurate ultrasound technique for evaluating right ventricular function.Measurement method:The sample volume was applied to the free wall of the RV and the peak velocity of tricuspid annulus motion was measured in the four-chamber section of the apex by tissue doppler imaging (TDI)
Right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) | at the time of 48 hours after enrollment
  RVEDA/LVEDA a simple and repeatable ultrasound method for evaluating dynamics changes of RV function.Methods: The RV end-diastolic area (RVEDA) and left ventricular(LV) end-systolic area (LVEDA) were measured on the apical four-chamber section by two-dimensional ultrasound
Pulmonary circulatory resistance (PVR) | at the time of 48 hours after enrollment
  Increased PVR can lead to deterioration of RV function.Pulse Doppler imaging (PWD) was used to obtain the pulmonary artery flow spectrum from the pulmonic valve on the short axial section of the parasternal great vessels.
Sequential Organ Failure Assessment score | at the time of 48 hours after enrollment
  The higher the Sequential Organ Failure Assessment(SOFA) score, the higher the disease risk factor and the higher the mortality rate(The highest score is 24, while the lowest score is 0).
cardiac index(CI) patients | at the time of 48 hours after enrollment
  CI is an important parameter to reflect the cardiac function of
Central venous oxygen saturation(ScvO2) | at the time of 48 hours after enrollment
  The patient's blood was collected through a central venous catheter for blood gas analysis to calculate SCVO2 to indicate tissue perfusion
systemic vascular resistance(SVR) | at the time of 48 hours after enrollment
  Peripheral vascular resistance is an important indicator of hemodynamics. It is not only a parameter reflecting cardiac afterload, but also a quantitative indicator reflecting the degree of patency of cerebrovascular microcirculation.
Mean arterial pressure (MAP) | at the time of 48 hours after enrollment
  MAP represents peripheral organ perfusion pressure.
Central venous pressure(CVP) | at the time of 48 hours after enrollment
  CVP is the pressure of the upper and lower vena cava entering the right atrium, measured by the upper and lower vena cava or the internal tube of the right atrium, which reflects the pressure of the right atrium, and is one of the main indicators for clinical observation of hemodynamics
systemic vascular resistance index(SVRI) | at the time of 48 hours after enrollment
  SVRI=80*(MAP-CVP)/CI
28-day mortality | Day 28 after study entry
  28-day mortality after study entry
in-hospital mortality | From the day patients admitted to hospital to the day death or discharge(up to 90 days)
  Any death occurred during hospitalization(up to 90 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

DOCUMENTS (1):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT05768230/Prot_000.pdf